CLINICAL TRIAL: NCT05546008
Title: Comparison Between Multislice CT 128 and Echocardiography in Diagnosis of Pediatric Congenital Heart Disease
Brief Title: Comparison Between Multislice CT and Echocardiography in Diagnosis of Pediatric Congenital Heart Disease
Acronym: CHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bahaa, DR, Assiut University
Other Study IDs: comparison between CT and Echo
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Multislice CT — all patient will be subjected to echocardigraphy and multislice ct and compare thier results
  Other Names: Echocardiography

SUMMARY:
1. Assesment of pediatric CHD by Echocardiography and Multislice CT before operation and compare with surgical results.
2. Compare echocardiogram and 128-Multislice spiral computed tomography(MSCT) in the diagnosis of pediatric CHD.
3. Confirm echocardiographic finding in pediatric CHD by(MSCT) and to show the role of MSCT in diagnosing of extra-cardia anomalies.
4. to show the role of MSCT as a useful tool in defintive diagnosis of congenital heart disease before operations which assist surgeons

DETAILED DESCRIPTION:
Congenital heart defect , also known as a congenital heart anomaly and congenital heart disease, is a defect in the structure of the heart or great vessels that is present at birth(1).

(congenital heart disease)(CHD), is the most frequent type of congenital birth deficiency disorder, with an incidence of 8% among newborns (2).

ECHO is the criterion standard and first-line diagnostic technique in diagnosing patients with CHD(11). For example, fetal echocardiography plays an important role in classifying the CHD in utero, allowing patients to be classified as having major, minor, or no CHD based on the echocardiographic results(3).

MSCT provides detailed, minimally invasive diagnosis and data on coronary artery anatomy in infants, children, and adults with CHD(13). CT,including CT angiography(CTA),is important in the evaluation of pediatric CHD.It can be used for accurate determination of complex cardiovascular anatomic features both before and after surgery and of a variety of post-treatment complications.

CT facilitate the assessment of extra-cardiac systemic and pulmonary arterial and venous structures(4).

Although the role of CT in the evaluation of pediatric congenital heart disease is being redefined and expanded, there are several generally accepted clinical indications for which the benefits of imaging outweigh the risks.First, CT can be used to evaluate patients with CHD known or suspected on the basis of echocardiographic findings for which further imaging is needed to characterize extra-cardiac anomalies before intervention.

The pulmonary arteries,pulmonary viens,and aortic arch and great vessels may be inadequately characterized at echocardiography, necessitating further assessment with CT (5).

History taking with emphasis on: age, gender, symptoms of heart failure as difficult breathing, palpitation, body swelling, and age of onset of these symptoms, as well as, syncopal attacks, cyanotic spills (blue color around lips), and failure to thrive.

2-Physical examination

1. Anthropometric measurement as weight,height,head circumference.
2. Vital signs as temperature,heart rate, respiratory rate,blood pressure.
3. General examination for detection of cyanosis and signs of heart failure as lower limb edema, hepatomegaly.
4. Cardiac examination for detection of pericardial bulge, dilated veins, abnormal pulsation,abnormal heart sounds and audible murmur.

3-Echocardiography ECHO will be performed using the Diamond Select iE33 Ultrasound system (Philips Medical Systems, Netherlands)(6). The procedures of the cardia acoustic window will be strictly followed. ECHO often will start with subcostal an acoustic window or subcostal acoustic window, and the major cardiovascular structures will be assessed according to Van Praagh segmental analysis(7).

4-128-MSCT Patients will be given oral chloral hydrate solution with a dosage of 50 mg/kg. The 64-MSCT examination will be performed by SOMATOM Perspective (Siemens, Germany)(8),with tube voltage of 80-100Kv, tube current of 80-100 mAs (vary during acquisition and according to the weight of the children), pitch of 1.2, and 0.6 mm collimation. A contrast medium dosage will be 1.2-2.0 mL/kg (Omnipaque 350 mg/mL), and will be followed by the same volume of saline chaser with an injection rate of 1-1.5 mL/s(9).

ELIGIBILITY:
Inclusion Criteria:

* children with congenital heart disease less than 18years

Exclusion Criteria:

* • Children with congenital heart disease >18 years.

  * Children suffering from renal disease .
  * Children with non-sinus rhythm .
  * Children who are allergic to iodinated contrast media .

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes
Study Population: children with congenital heart disease less than 18years
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
comparison between Multislice CT and Echo cardiography in diagnosis of congenital heart disease | baseline
  The study will be conducted at Assiut University Children Hospital from septemper 2022 to septemper 2023 on children with congenital heart disease
  1-Echocardiography ECHO will be performed using the Diamond Select iE33 Ultrasound system (Philips Medical Systems, Netherlands)(6) 2-128-MSCT Patients will be given oral chloral hydrate solution with a dosage of 50 mg/kg. The 64-MSCT examination will be performed by SOMATOM Perspective

REFERENCES:
- [Background] VANPRAAGH R, VANPRAAGH S, VLAD P, KEITH JD. ANATOMIC TYPES OF CONGENITAL DEXTROCARDIA: DIAGNOSTIC AND EMBRYOLOGIC IMPLICATIONS. Am J Cardiol. 1964 Apr;13:510-31. doi: 10.1016/0002-9149(64)90159-6. No abstract available. PMID 14136294
- [Background] Alakhfash AA, Tamimi OR, Al-Khattabi AM, Najm HK. Treatment options for transposition of the great arteries with ventricular septal defect complicated by pulmonary vascular obstructive disease. J Saudi Heart Assoc. 2009 Jul;21(3):187-90. doi: 10.1016/j.jsha.2009.06.008. Epub 2009 Aug 5. PMID 23960571
- [Background] Pasquini L, Sanders SP, Parness I, Colan S, Keane JF, Mayer JE Jr, Kratz C, Foran RB, Marino B, Van Praagh S, et al. Echocardiographic and anatomic findings in atrioventricular discordance with ventriculoarterial concordance. Am J Cardiol. 1988 Dec 1;62(17):1256-62. doi: 10.1016/0002-9149(88)90270-6. PMID 3195487
- [Background] Wang XM, Wu LB, Sun C, Liu C, Chao BT, Han B, Zhang YT, Chen HS, Li ZJ. Clinical application of 64-slice spiral CT in the diagnosis of the Tetralogy of Fallot. Eur J Radiol. 2007 Nov;64(2):296-301. doi: 10.1016/j.ejrad.2007.02.026. Epub 2007 Mar 30. PMID 17399932
- [Background] Liu H, Juan YH, Chen J, Xie Z, Wang Q, Zhang X, Liang C, Huang H, Kwong RY, Saboo SS. Anomalous Origin of One Pulmonary Artery Branch From the Aorta: Role of MDCT Angiography. AJR Am J Roentgenol. 2015 May;204(5):979-87. doi: 10.2214/AJR.14.12730. PMID 25905931
- [Background] Watts JR Jr, Sonavane SK, Nath PH, Singh SP. Pictorial review of the role of multidetector computed tomography imaging in the postoperative evaluation of congenital heart disease. Curr Probl Diagn Radiol. 2014 Jul-Aug;43(4):205-18. doi: 10.1067/j.cpradiol.2014.04.001. PMID 24948213